CLINICAL TRIAL: NCT06827171
Title: Impact of Low-level Laser and Aerobic Exercise on Peripheral Arterial Outcomes in Patients With Type 2 Diabetes
Brief Title: Impact of LLL and Aerobic Exercise on Peripheral Arterial Outcomes in Patients With Type 2 Diabetes
Acronym: LLLT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nouran Hesham Slama Younis (Other)
Responsible Party: Sponsor-Investigator, Nouran Hesham Slama Younis, Clinical investigator, police hospital, Egypt, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: P.T.REC/012/004935
Record Dates: First submitted 2025-01-19; First posted 2025-02-14 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Peripheral artery Disease; Low level laser; Aerobic exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Peripheral Arterial Disease | interventions — Exercise; Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: the study is going to contain 2 experimental groups, the first one will receive combined therapy (aerobic exercise program for PAD + low-level laser therapy) the other group will receive aerobic exercise program for PAD only.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Study group A: Aerobic exercise+ low-level Laser therapy (Experimental): (Study group A): It will receive a low-level laser (scanning laser) on the course of the posterior tibial and anterior tibial artery combined with an aerobic exercise program for peripheral artery disorder for 12 weeks (3 sessions/ week).
  Interventions: Combination Product: aerobic exercise + low-level laser therapy; Other: Aerobic exercise
- Control group B: Aerobic Exercise group B (Experimental): group B: They will receive aerobic exercise for 12 weeks. aerobic exercise program for peripheral arterial disorders and intermittent claudication.
  Interventions: Other: Aerobic exercise

INTERVENTIONS:
Combination Product: aerobic exercise + low-level laser therapy — low- level laser parameters: The wavelength: 808 +/- 5nm The power: output is 450 Mw Type of beam: red laser beam. Beam Divergent >,025 rad+/- ,005rad Nominal Distance of Sight hazard >8m The duration: is 20 min for each artery. Treatment period: 3 times/week for 3 months.
  Arms: Study group A: Aerobic exercise+ low-level Laser therapy
Other: Aerobic exercise — Aerobic exercise Frequency = 3sessions/week duration: 10 min warm up and 10 min cool down/ 30 min stance phase Intensity: moderate intensity initiating with 50% HR max to end 75% HR max

SUMMARY:
Diabetes is one of the fastest-growing diseases worldwide, It has Devastating macrovascular complications (cardiovascular disease) and microvascular complications (such as diabetic kidney disease, diabetic retinopathy, and neuropathy) In Egypt, factors in patients that affect diabetic control include the patient's education and occupation and smoking status. Physical exercise is important for diabetes control. Metformin and investigation availability have a positive association with diabetes control.

Diabetes mellitus increases the risk and accelerates the course of peripheral artery disease, making patients more susceptible to ischemic events and infections and delaying tissue healing. The current understanding of pathogenic mechanisms is mainly based on the negative influence of diabetes mellitus on atherosclerotic disease and inflammation (Fadini et al., 2020).) An early diagnosis of peripheral arterial diseases PAD and correctly identifying patients with Chronic limb-threatening ischemia CLTI are crucial in patients with diabetes to improve outcomes.

Several treatment strategies can be subdivided into lifestyle modification, medical management, endovascular therapies, and surgical interventions for the treatment of PAD.

Exercise training improves walking ability, distances, physical function, and vitality. Physical activity by supervised exercise is recommended in first-line therapy for intermittent claudication by SVS, ESVS, and AHA (Treat-Jacobson et al., 219) More specifically, a supervised exercise program consists of walking a minimum of three times per week (30-60 min/session) for at least 12 weeks Therapeutic laser treatment, also known as low-level laser therapy (LLLT), offers numerous benefits. It is non-surgical, promotes tissue healing, and reduces edema, inflammation, and pain.

DETAILED DESCRIPTION:
The participants will be submitted into two equal groups in numbers:

Group A (Study group) n=20 will receive a low-level laser (scanning laser) combined with an aerobic exercise program for 12 weeks (3 sessions/ week).

Group B (control group) n=20: Who will receive aerobic exercise for 12 weeks (3sessions/week) All patients with their prescribed medications (hypoglycemic, antiplatelet, anticoagulants, antihypertensive, vasodilators, analgesics)

ELIGIBILITY:
Inclusion Criteria:

* Their ages will range from 55- 65 years, for both genders.
* Body Mass Index of 25-29.9kg/m2.
* Glycated hemoglobin (HbA1c) from 7 to 9 %.
* The patient has suffered from diabetes for more than 5 years.
* Patient with mild to moderate PAD on Rutherford classification stages (1-3)

Exclusion Criteria:

1. Patients with a history of hypo-hyperglycemic coma.
2. Uncontrolled cardiovascular complications, and ischemic heart disease.
3. Photosensitivity, Malignancy, Anemia, Hemorrhagic diseases (contraindication to laser)
4. Deep venous thrombosis, acute thromboses.
5. Cerebrovascular disease.
6. Patients with Monckeberg sclerosis.
7. Patient with resting pain critical limb ischemia, diabetic foot, and peripheral edema, asymptomatic PAD, Diabetic neuropathy.
8. Patient with minor/ or major amputations.
9. A patient with positive smoking

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
body mass index | 3 month
  Body mass index (Kg/M^2): by dividing the weight by kilogram over Height by meter square.
peak systolic velocities (PSV) | 3 months
  Duplex ultrasonography of the lower extremity arteries, from common femoral to pedal arteries is used to measure PSV
  * Peak systolic velocities (PSV) were recorded in meters per second (Ugwu et al., 2021).
  * The normal peak systolic velocity (PSV) in peripheral lower limb arteries varies from 45-180 cm/s (Abdelrahman, 2010).
  Severe arterial disease manifests as a PSV over 200 cm/s, monophasic waveform, and spectral broadening of the Doppler waveform.
Ankle-Brachial Index (ABI) % | 3 months
  • Ankle-Brachial Index (ABI) is a ratio of the highest ankle systolic blood pressure obtained in the anterior tibial/ dorsalis pedis or posterior tibial artery to that of the highest brachial systolic pressure.
  An ABI < 0.9 was diagnostic of PAD and values were stratified according to severity as:
  * 0.7-0.89 = mild arterial obstruction.
  * 0.5-0.69 = moderate arterial obstruction.
  * ≤ 0.5 = severe arterial obstruction.
The visual analog scale (VAS) questionnaire for pain | 3 months
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." Delgado etal., 2018).
  * no pain (0-4 mm)
  * mild pain(5-44 mm)
  * moderate pain (45-74 mm)
  * severe pain (75-100 mm). (Weigl K et al., 2021)
The Edinburgh Claudication Questionnaire (ECQ) | 3 months
  The Edinburgh Claudication Questionnaire (ECQ) Definition of positive classification requires all of the following responses: \Yes" to (1), \No" to (2), \Yes" to (3), Grade 1 \No" to (4), and Grade 2 \Yes" to (4). If these criteria are met, a typical claudicant is one who indicates the pain is in the calf, regardless of whether the pain is also marked at other sites; a diagnosis of atypical claudication is made when the pain is marked in the thigh or buttock, in the absence of any calf pain. Subjects should not be diagnosed with claudication if the pain is indicated in the hamstrings, feet, shins, and joints, or radiates in the absence of any calf pain

SECONDARY OUTCOMES:
The initial claudication distance and The absolute claudication distance (meters) | 3 months
  The initial claudication distance (ICD), or pain-free walking distance; is the distance walked at the onset of claudication pain The absolute claudication distance (ACD), or maximal walking distance at which claudication pain becomes so severe that the patient is forced to stop (Jongert et al., 2003)
Maximum oxygen consumption Vo^2 max ((ml/kg/min)) | 3 months
  depend on Modified Bruce protocol with the treadmill. Modified Bruce protocol, the first stage at 1.7mph and 0% grade second stage at 1.7 mph 5% grade, and the third stage at 1.7 mph and 10% grade.
  The test score is the time taken on the test, in minutes. This can also be converted to an estimated VO2 max score using the calculator below and the following formulas, where the value "T" is the total time completed (expressed in minutes and fractions of a minute e.g. 9 minutes 25 seconds = 9.25 minutes).
  Men : VO2max (ml/kg/min) = 14.76 -(1.379 × T) + (0.451 × T²)-(0.012 × T³) Women: VO2max (ml/kg/min) = 4.38x T -3.9 (ACSM, 2023)

CONTACTS AND LOCATIONS:
Overall Officials: Nesreen Gh EL NAHAS, doctor, Principal Investigator — head of physical therapy department for internal medicine, Cairo university.
Locations (1):
- Cairo University, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No